CLINICAL TRIAL: NCT05324254
Title: Effect of Weighted Blankets on Perioperative Anxiety and Postsurgical Pain
Brief Title: Weighted Blankets for Postsurgical Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Laura Case, Adjunct Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 210487
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postsurgical
Keywords: mastectomy; anxiety; blankets
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Partial masking: Although blanket heaviness will be perceived, blanket weights tested in the study will not be disclosed to participants. Wait-list control group will know they are not receiving active intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heavier blanket (Experimental): A heavier blanket will be worn overnight for 3 months. Blanket weight cannot be disclosed without unblinding participants.
  Interventions: Device: Weighted blanket
- Lighter blanket (Experimental): A lighter blanket will be worn overnight for 3 months. Blanket weight cannot be disclosed without unblinding participants.
  Interventions: Device: Weighted blanket
- Waitlist control (No Intervention): No blanket will be provided until the end of the study; participants will sleep with their normal bedding.

INTERVENTIONS:
Device: Weighted blanket — A weighted blanket is a blanket with extra weight sewn in for added pressure to the body.
  Arms: Heavier blanket; Lighter blanket

SUMMARY:
The strongest psychological predictor of persistent pain after surgery is anxiety before surgery. The weight of blanket a person uses overnight may alter both anxiety and pain levels. The proposed study will determine whether a heavier or lighter blanket alters presurgical anxiety or postsurgical pain in individuals undergoing a breast surgery. We will also study whether any blanket-induced changes in postsurgical pain are related to reductions in anxiety before surgery induced by the blanket. Finally, we will examine clinical and psychological factors that might explain differences in how surgical patients respond to blanket weight. This research will improve our understanding of whether blanket weight can alter anxiety before a surgery or pain after a surgery.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Undergoing breast surgery
* Willing to sleep with a weighted blanket for up to 3 months
* BMI of at least 18.5 and able to safely lift up to 15lb
* Willing and able to use their personal smartphone for the ecological momentary assessment app to submit ratings using personal data plan

Exclusion Criteria:

* Pregnancy
* Chronic high-dose opioid use
* Current or previous use of a weighted blanket
* Claustrophobia
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety ratings from before to during blanket use before surgery | arrival to surgical center and final rating prior to surgery
  Anxiety ratings will be compared before and during use of weighted blanket on the following scale: "Extremely anxious" to "Neutral" to "Extremely calm"
Change in postsurgical pain from before to after overnight blanket use | baseline (before surgery) and 1 and 3 months after surgery
  Brief Pain Inventory score will be compared before and after overnight use of assigned blanket
Change in medication use from before to after overnight blanket use | baseline (before surgery) and 1 and 3 months after surgery
  Medications taken in past 24 hours will be self-reported

SECONDARY OUTCOMES:
Change in postsurgical pain from before to after overnight blanket use | baseline, 1 week, 1 month, and 3 months
  Pain ratings will be compared before and after overnight use of assigned blanket: Pain Intensity visual analog scale "No pain" to "Most intense pain imaginable" and Pain unpleasantness visual analog scale: "No unpleasantness" to "Most unpleasant pain imaginable"
Change in medication use from before to after overnight blanket use | baseline, 1 week, 1 month, and 3 months
  Medications taken in past 24 hours will be self-reported

CONTACTS AND LOCATIONS:
Locations (1):
- Actri, Ucsd, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No